CLINICAL TRIAL: NCT05871632
Title: The China CardioMyopathy Registry Study
Acronym: CHINA-CM
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lei.Song,MD.&ph.D, Principal Investigator, Clinical Professor, China National Center for Cardiovascular Diseases
Other Study IDs: CHINA-CM
Record Dates: First submitted 2023-05-10; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiomyopathy is the most common inherited cardiovascular disease, showing family aggregation, so it has a huge psychological and economic burden on family members. Studying the clinical characteristics of patients with cardiomyopathy is helpful for further diagnosis, treatment and management, which has important clinical and social significance.

DETAILED DESCRIPTION:
In this study, patients hospitalized with cardiomyopathy as the primary discharge diagnosis in China are recruited prospectively after informed consent was given. The investigator will collect the baseline clinical characteristics of the patients at enrollment, including comprehensive physical examination, laboratory testing of blood and urine, electrocardiography, 24-hour Holter, echocardiography, MRI and other examinations if necessary. Data are collected with the use of case report forms (CRFs) and are entered into a web-based system. A 6 mL venous blood sample is obtained from consenting patients. Each participant is scheduled to be followed up by telephone every 12 months after admission to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary discharge diagnosis meeting one of the following subtypes of cardiomyopathy were enrolled, including HCM, DCM, ACM, RCM, left ventricular non-compaction, cardiac amyloidosis, Fabry disease, Pompe disease, Danon disease, and PRKAG2 cardiac syndrome.

Exclusion Criteria:

* Patients who refuse to sign the informed consent or decline follow-up.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized with cardiomyopathy as the primary discharge diagnosis are recruited prospectively from multiple centers in China between July 1, 2023 and June 30, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
number of participants with cardiovascular deaths | an average of 1 year
  including sudden cardiac death and deaths due to heart failure and stroke

SECONDARY OUTCOMES:
number of participants with heart failure | an average of 1 year
  progress to level III or IV in New York Heart Association class
number of participants with stroke | an average of 1 year
  including cerebral infraction and hemorrhage
number of participants with myocardial infarction | an average of 1 year
  including ST-segment elevation myocardial infarction and non-ST-segment elevation myocardial infarction
number of participants with all-cause deaths | an average of 1 year
  including deaths due to any causes

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided